CLINICAL TRIAL: NCT02616562
Title: A Randomised, Multinational, Active-controlled, (Open-labelled), Dose Finding, (Double-blinded), Parallel Group Trial Investigating Efficacy and Safety of Once-weekly NNC0195-0092 Treatment Compared to Daily Growth Hormone Treatment (Norditropin® FlexPro®) in Growth Hormone Treatment naïve Pre-pubertal Children With Growth Hormone Deficiency
Brief Title: Investigating Efficacy and Safety of Once-weekly NNC0195-0092 Treatment Compared to Daily Growth Hormone Treatment (Norditropin® FlexPro®) in Growth Hormone Treatment naïve Pre-pubertal Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8640-4172; 2015-000531-32 (EudraCT Number); U1111-1166-7062 (Other: WHO)
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children
MeSH Terms: interventions — somapacitan; NNC0195-0092

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort I Norditropin/somapacitan (Experimental): Participants received Norditropin subcutaneously daily in main trial period, extension trial period and safety extension trial period. After completing the safety extension trial period (week 156), participants who received Norditropin were allocated to open-labelled Somapacitan dose 3 subcutaneously once weekly for the 208-week (up till week 364) long-term safety extension period. After week 364, participants received somapacitan dose 3 subcutaneously once weekly until somapacitan was available for prescription for children with GHD in their country or until August 2024, at the latest.
  Interventions: Drug: somapacitan; Drug: Norditropin® FlexPro® pen
- Cohort I somapacitan pooled (Experimental): Participants were randomized (1:1:1) to receive Somapacitan treatment (dose 1/dose 2/dose 3) subcutaneously once-weekly during the 26-week main trial period and the 26-week extension trial period. After completing the main and extension trial periods (week 52), all participants initially randomized to double-blinded Somapacitan received open-labelled Somapacitan dose 3 for the 104-week safety extension trial period. After completing the safety extension trial period (week 156), all participants in cohort I were allocated to open-labelled somapacitan dose 3 for the 208-week (up till week 364) long-term safety extension period. In extension after week 364 period participants received somapacitan dose 3 subcutaneously once weekly until somapacitan was available for prescription for children with GHD in their country or until August 2024, at the latest.
  Interventions: Drug: somapacitan
- Cohort II somapacitan previously treated (Experimental): Participant who was previously treated with GH (Growth hormone) prior to enrollment in the trial at week 156, received somapacitan dose 3 subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
  Interventions: Drug: somapacitan
- Cohort III somapacitan treatment naive (Experimental): Participants who were naive to treatment with GH prior to enrolment in the trial at week 156, received open-labelled somapacitan dose 3 subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
  Interventions: Drug: somapacitan
- Cohort III somapacitan previously treated (Experimental): Participants who were previously treated with GH prior to enrollment in the trial at week 156, received open-labelled somapacitan dose 3 subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
  Interventions: Drug: somapacitan

INTERVENTIONS:
Drug: somapacitan — Administered subcutaneously (s.c., under the skin) once-weekly.
  Other Names: NNC0195-0092
Drug: Norditropin® FlexPro® pen — Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Cohort I Norditropin/somapacitan

SUMMARY:
This trial is conducted globally. The aim of the trial is to investigate efficacy and safety of once-weekly NNC0195-0092 treatment compared to daily growth hormone treatment (Norditropin® FlexPro®) in growth hormone treatment naïve pre-pubertal children with growth hormone deficiency.

The main trial period will consist of 26 weeks of treatment, followed by a 26 week extension period.

ELIGIBILITY:
Inclusion Criteria:

* Boys: Tanner stage 1 for pubic hair and testis volume below 4 ml , age at least 2 years and 26 weeks and below or equal to 10.0 years at screening
* Girls: Tanner stage 1 for breast development (no palpable glandular breast tissue) and pubic hair, age at least 2 years and 26 weeks and below or equal to 9.0 years at screening
* Confirmed diagnosis of GHD (growth hormone deficiency) within 12 months prior to screening as determined by two different GH (growth hormone) stimulation tests, defined as a peak GH level of below or equal to 7.0 ng/ml. For children with three or more pituitary hormone deficiencies only one GH stimulation test is needed
* No prior exposure to GH therapy and/or IGF-I (insulin-like growth factor I) treatment
* Height of at least 2.0 standard deviations below the mean height for chronological age (CA) and gender according to the standards of Centers for Disease Control and Prevention 2-20 years: Girls/Boys stature-for-age and weight-for-age percentiles CDC at screening
* Annualized height velocity (HV) below the 25th percentile for CA (chronological age) and gender or below -0.7 SD (standard deviation) score for CA and sex, according to the standards of Prader calculated over a time span of minimum 6 months and maximum 18 months

Exclusion Criteria:

* Any clinically significant abnormality likely to affect growth or the ability to evaluate
* growth with standing measurements: Chromosomal aneuploidy and significant gene mutations causing medical "syndromes" with short stature, including but not limited to Turner syndrome, Laron syndrome, Noonan syndrome, or absence of GH receptors. Congenital abnormalities (causing skeletal abnormalities), including but not limited to Russell-Silver Syndrome, skeletal dysplasias. Significant spinal abnormalities including but not limited to scoliosis, kyphosis and spina bifida variants
* Children born small for gestational age (SGA - birth weight and/or birth length below-2 SD for gestational age)
* Concomitant administration of other treatments that may have an effect on growth, including but not limited to methylphenidate for treatment of attention deficit hyperactivity disorder (ADHD)
* Prior history or presence of malignancy and/or intracranial tumour

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (89):
- United States (27):
  - Children's of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Novo Nordisk Clinical Trial Call Center, San Diego, California
  - The Regents of the Univ of CA, San Diego, California
  - Rocky Mt Ped and Endo, Centennial, Colorado
  - Ped Endo Assoc PC-G.V, Greenwood Village, Colorado
  - Nemours/AI duPont Hosp-Chld, Wilmington, Delaware
  - The Endocrine Center, Pembroke Pines, Florida
  - Childrens Hospital of Chicago, Chicago, Illinois
  - Riley Hospital For Children, Indianapolis, Indiana
  - Novo Nordisk Clinical Trial Call Center, Minneapolis, Minnesota
  - University of Minnesota_Minneapolis_2, Minneapolis, Minnesota
  - Goryeb Children's Hospital, Morristown, New Jersey
  - Novo Nordisk Clinical Trial Call Center, Morristown, New Jersey
  - Rutgers-Rwjms, New Brunswick, New Jersey
  - UBMD Peds-Div of Endo/Diabetes, Buffalo, New York
  - Novo Nordisk Clinical Trial Call Center, Mineola, New York
  - NYU Langone Hospital-LI, Mineola, New York
  - CCHMC_Cinc, Cincinnati, Ohio
  - Novo Nordisk Clinical Trial Call Center, Cincinnati, Ohio
  - University Of Oklahoma-Tulsa, Tulsa, Oklahoma
  - Dell Pediatric Research Institute, Austin, Texas
  - Endocrine Associates Of Dallas, Plano, Texas
  - Children's Hsptl Of The Kings, Norfolk, Virginia
  - MultiCare Inst for Res & Innov, Tacoma, Washington
- Austria (7):
  - Kepler Universitätsklinikum GmbH - Med Campus IV (vorm.LFKK), Linz, Upper Austria
  - Med. Univ. Graz -Klinische Abteilung f. Allgemeine Pädiatrie, Graz
  - Graz
  - LKH Salzburg- Univ. Klinik f. Kinder- und Jugendheilkunde, Salzburg
  - LKH St. Poelten, Kinder-und Jugendheilkunde, Sankt Pölten
  - Landeskrankenhaus Villach, Villach
  - Salzkammergut-Klinikum Vöcklabruck, Vöcklabruck
- Belgium (5):
  - UZ Brussel, Brussels
  - Brussels
  - Cliniques Universitaires Saint-Luc - Serv. Pédiatrie, Brussels
  - UZ Leuven - Kindergeneeskunde, Leuven
  - CHU de Liège, site N.-D. des Bruyères, Liège
- Brazil (4):
  - Serviço de Endocrinologia e Metabologia do HC-UFPR, Curitiba, Paraná
  - Hospital São Lucas - PUC/RS, Porto Alegre, Rio Grande do Sul
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - São Paulo, São Paulo
- The Hospital for Sick Children, Toronto, Ontario, Canada
- France (7):
  - Centre Hospitalier Universitaire D'Angers-2, Angers
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Pellegrin, Bordeaux
  - Bordeaux
  - Centre Hospitalier Universitaire de Nantes-Hopital Enfant-Adolescent, Nantes
  - Ap-Hp-Hopital Necker, Paris
  - HOPITAL SUD de RENNES, Rennes
  - HOPITAL DES ENFANTS-HOPITAL PAULE DE VIGUIER - Pharmacie, Toulouse
- Germany (3):
  - Frankfurt
  - Endokrinologikum Frankfurt, Frankfurt am Main
  - Uniklinik Ulm - Dt. Zentrum für Kinder- und Jugendgesundheit (DZKJ), Ulm
- India (4):
  - Amrita Institute Of Medical Sciences & Research Centre, Kochi, Kerala
  - Jehangir Clinical Development Centre, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Dehli, New Delhi
  - New Dehli, New Delhi
- Israel (6):
  - Soroka MC - Pediatric Endocrinology, Beersheba
  - Rambam MC - Department of Pediatrics A, Haifa
  - Meir MC - Department of Paediatrics, Kfar Saba
  - Kfar Saba
  - Schneider MC - Endrocrinology and Diabetes, Petah Tikva
  - Sheba MC - Pediatric endocrinology and adolescent diabetes clinics, Tel Litwinsky
- Japan (11):
  - Kyushu Univ. HP, Maternity & Perinatal Care Center, Fukuoka
  - Kurume University Hospital, Pediatrics, Fukuoka
  - St. Marianna University School of Medicine Hospital_Pediatrics, Kanagawa
  - Univ.HP, Kyoto Pref Univ of Medicine, Dept. of Pediatrics, Kyoto
  - Osaka City General Hospital, Pediatric Endocrinology and Me, Osaka
  - JCHO Osaka Hospital_Pediatric, Osaka
  - Osaka Women's and Children's Hospital, Osaka
  - Institute of Science Tokyo Hospital_Pediatrics, Tokyo
  - Tokyo Medical and Dental University Hospital, Tokyo
  - National Center for Child Health and Dev, Endo and Metabo, Tokyo
  - Tokyo
- Slovenia (2):
  - University Children's Hospital, Ljubljana
  - Ljubljana
- Sweden (3):
  - Astrid Lindgrens Barnsjukhus, Stockholm
  - Stockholm
  - Barn och ungdomscentrum Västerbotten, Umeå
- Turkey (Türkiye) (6):
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi, Adana
  - Hacettepe Üniversitesi Hastanesi- Endokrinoloji, Ankara
  - I.U Istanbul Medical Faculty, Istanbul
  - Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Marmara Üniversitesi Pendik EAH- Başıbüyük Yerleşkesi- Kardiyoloji, Istanbul
- Ukraine (3):
  - Ivano-Frankivsk Regional Clinical Children Hospital - Endocrinology dept., Ivano-Frankivsk
  - Kiev
  - Komisarenko Institute of Endocrinology and Metabolism of NAMSU - Department of paediatric endocrine pathology, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Savendahl L, Battelino T, Hojby Rasmussen M, Brod M, Rohrich S, Saenger P, Horikawa R. Weekly Somapacitan in GH Deficiency: 4-Year Efficacy, Safety, and Treatment/Disease Burden Results From REAL 3. J Clin Endocrinol Metab. 2023 Sep 18;108(10):2569-2578. doi: 10.1210/clinem/dgad183. PMID 36995872
- [Derived] Savendahl L, Battelino T, Hojby Rasmussen M, Brod M, Saenger P, Horikawa R. Effective GH Replacement With Once-weekly Somapacitan vs Daily GH in Children with GHD: 3-year Results From REAL 3. J Clin Endocrinol Metab. 2022 Apr 19;107(5):1357-1367. doi: 10.1210/clinem/dgab928. PMID 34964458
- [Derived] Savendahl L, Battelino T, Brod M, Hojby Rasmussen M, Horikawa R, Juul RV, Saenger P; REAL 3 study group. Once-Weekly Somapacitan vs Daily GH in Children With GH Deficiency: Results From a Randomized Phase 2 Trial. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1847-61. doi: 10.1210/clinem/dgz310. PMID 31917835
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 30 sites in 11 countries.
Pre-assignment Details: The study has 3 cohorts. Cohort I participants were randomised (1:1:1:1) to receive norditropin/somapacitan(0.04/0.08/0.16 mg/kg) until week 52. After week 52, participants who were randomised to somapacitan were allocated to open labelled somapacitan and those who randomised to norditropin received same treatment. After week 156, all cohort I participants received somapacitan until August 24.
  Participants in cohorts II and III were given somapacitan from enrolment (week 156) until August 24.
Groups:
- Main - Cohort I Norditropin 0.034 mg/kg: Participants received norditropin 0.034 milligram per kilogram (mg/kg) subcutaneously daily during (26 week) main trial period.
- Main - Cohort I Somapacitan 0.04 mg/kg: Participants received somapacitan 0.04 mg/kg subcutaneously once-weekly during the (26 week) main trial period.
- Main - Cohort I Somapacitan 0.08 mg/kg: Participants received somapacitan 0.08 mg/kg subcutaneously once- weekly during (26 week) main trial period.
- Main - Cohort Somapacitan 0.16 mg/kg: Participants received somapacitan 0.16 mg/kg subcutaneously once- weekly during (26 week) main trial period.
- Extension - Cohort I Norditropin 0.034 mg/kg: Participants received norditropin 0.034 mg/kg subcutaneously daily during (26 week) extension trial period.
- Extension - Cohort I Somapacitan 0.04 mg/kg: Participants received 0.04 mg/kg subcutaneously once-weekly during the (26 week) extension trial period.
- Extension - Cohort I Somapacitan 0.08 mg/kg: Participants received 0.08 mg/kg subcutaneously once-weekly during the (26 week) extension trial period.
- Extension - Cohort I Somapacitan 0.16 mg/kg: Participants received 0.16 mg/kg subcutaneously once-weekly during the (26 week) extension trial period.
- Safety Extension - Cohort I Norditropin 0.034 mg/kg: Participants randomised to norditropin 0.034 mg/kg continued same treatment subcutaneously daily during (104 week) safety extension period.
- Safety Extension - Cohort I Somapacitan 0.16 mg/kg: Participants initially randomized to double-blinded somapacitan treatment (0.04/0.08/0.16 mg/kg) during main and extension period received open-labelled somapacitan 0.16 mg/kg subcutaneously once-weekly during 104 week safety extension period.
- Long Term Safety Extension - Cohort I Norditropin/Somapacitan: Participants who received norditropin until week 156 were given somapacitan 0.16 mg/kg subcutaneously once weekly for the 208-week long term safety extension period (up till week 364)
- Long Term Safety Extension - Cohort I Somapacitan 0.16 mg/kg: Participants received somapacitan 0.16 mg/kg subcutaneously once weekly for the 208-week long term safety extension period (up till week 364)
- Long Term Safety Extension - Cohort II Somapacitan Previously Treated: Participant who was previously treated with GH (Growth hormone) prior to enrollment in the trial at week 156, received somapacitan 0.16 mg/kg subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
- Long Term Safety Extension - Cohort III Somapacitan Treatment Naive: Participants who were naive to treatment with GH prior to enrollment in the trial at week 156, received open-labelled somapacitan 0.16 mg/kg subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
- Long Term Safety Extension - Cohort III Somapacitan Previously Treated: Participants who were previously treated with GH prior to enrollment in the trial at week 156, received open-labelled somapacitan 0.16 mg/kg subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
- Extension After Week 364 - Cohort I Norditropin/Somapacitan; Extension After Week 364 - Cohort I Somapacitan 0.16 mg/kg: Participants received somapacitan 0.16 mg/kg subcutaneously once weekly until somapacitan was available for prescription for children with GHD in their country or until August 2024, at the latest.
Period: Main Period (26 Weeks)
Arm/Group | Main - Cohort I Norditropin 0.034 mg/kg | Main - Cohort I Somapacitan 0.04 mg/kg | Main - Cohort I Somapacitan 0.08 mg/kg | Main - Cohort Somapacitan 0.16 mg/kg | Extension - Cohort I Norditropin 0.034 mg/kg | Extension - Cohort I Somapacitan 0.04 mg/kg | Extension - Cohort I Somapacitan 0.08 mg/kg | Extension - Cohort I Somapacitan 0.16 mg/kg | Safety Extension - Cohort I Norditropin 0.034 mg/kg | Safety Extension - Cohort I Somapacitan 0.16 mg/kg | Long Term Safety Extension - Cohort I Norditropin/Somapacitan | Long Term Safety Extension - Cohort I Somapacitan 0.16 mg/kg | Long Term Safety Extension - Cohort II Somapacitan Previously Treated | Long Term Safety Extension - Cohort III Somapacitan Treatment Naive | Long Term Safety Extension - Cohort III Somapacitan Previously Treated | Extension After Week 364 - Cohort I Norditropin/Somapacitan | Extension After Week 364 - Cohort I Somapacitan 0.16 mg/kg
Started | 14 | 16 | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 14 | 15 | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension Period (26 Weeks)
Arm/Group | Main - Cohort I Norditropin 0.034 mg/kg | Main - Cohort I Somapacitan 0.04 mg/kg | Main - Cohort I Somapacitan 0.08 mg/kg | Main - Cohort Somapacitan 0.16 mg/kg | Extension - Cohort I Norditropin 0.034 mg/kg | Extension - Cohort I Somapacitan 0.04 mg/kg | Extension - Cohort I Somapacitan 0.08 mg/kg | Extension - Cohort I Somapacitan 0.16 mg/kg | Safety Extension - Cohort I Norditropin 0.034 mg/kg | Safety Extension - Cohort I Somapacitan 0.16 mg/kg | Long Term Safety Extension - Cohort I Norditropin/Somapacitan | Long Term Safety Extension - Cohort I Somapacitan 0.16 mg/kg | Long Term Safety Extension - Cohort II Somapacitan Previously Treated | Long Term Safety Extension - Cohort III Somapacitan Treatment Naive | Long Term Safety Extension - Cohort III Somapacitan Previously Treated | Extension After Week 364 - Cohort I Norditropin/Somapacitan | Extension After Week 364 - Cohort I Somapacitan 0.16 mg/kg
Started | 0 | 0 | 0 | 0 | 14 | 15 | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 14 | 15 | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Safety Extension Period (104 Weeks)
Arm/Group | Main - Cohort I Norditropin 0.034 mg/kg | Main - Cohort I Somapacitan 0.04 mg/kg | Main - Cohort I Somapacitan 0.08 mg/kg | Main - Cohort Somapacitan 0.16 mg/kg | Extension - Cohort I Norditropin 0.034 mg/kg | Extension - Cohort I Somapacitan 0.04 mg/kg | Extension - Cohort I Somapacitan 0.08 mg/kg | Extension - Cohort I Somapacitan 0.16 mg/kg | Safety Extension - Cohort I Norditropin 0.034 mg/kg | Safety Extension - Cohort I Somapacitan 0.16 mg/kg | Long Term Safety Extension - Cohort I Norditropin/Somapacitan | Long Term Safety Extension - Cohort I Somapacitan 0.16 mg/kg | Long Term Safety Extension - Cohort II Somapacitan Previously Treated | Long Term Safety Extension - Cohort III Somapacitan Treatment Naive | Long Term Safety Extension - Cohort III Somapacitan Previously Treated | Extension After Week 364 - Cohort I Norditropin/Somapacitan | Extension After Week 364 - Cohort I Somapacitan 0.16 mg/kg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 41 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — treatment discontinued before visit 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Long Term Safety Extension (208 Weeks)
Arm/Group | Main - Cohort I Norditropin 0.034 mg/kg | Main - Cohort I Somapacitan 0.04 mg/kg | Main - Cohort I Somapacitan 0.08 mg/kg | Main - Cohort Somapacitan 0.16 mg/kg | Extension - Cohort I Norditropin 0.034 mg/kg | Extension - Cohort I Somapacitan 0.04 mg/kg | Extension - Cohort I Somapacitan 0.08 mg/kg | Extension - Cohort I Somapacitan 0.16 mg/kg | Safety Extension - Cohort I Norditropin 0.034 mg/kg | Safety Extension - Cohort I Somapacitan 0.16 mg/kg | Long Term Safety Extension - Cohort I Norditropin/Somapacitan | Long Term Safety Extension - Cohort I Somapacitan 0.16 mg/kg | Long Term Safety Extension - Cohort II Somapacitan Previously Treated | Long Term Safety Extension - Cohort III Somapacitan Treatment Naive | Long Term Safety Extension - Cohort III Somapacitan Previously Treated | Extension After Week 364 - Cohort I Norditropin/Somapacitan | Extension After Week 364 - Cohort I Somapacitan 0.16 mg/kg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 41 | 1 | 4 | 12 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 33 | 1 | 2 | 9 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 0 | 2 | 3 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Growth velocity in 9 months is 1 cm (1.3 CM/Y) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject was discontinued from trial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Principal Investigator's decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adult height reached | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Extension After Week 364 (78 Weeks)
Arm/Group | Main - Cohort I Norditropin 0.034 mg/kg | Main - Cohort I Somapacitan 0.04 mg/kg | Main - Cohort I Somapacitan 0.08 mg/kg | Main - Cohort Somapacitan 0.16 mg/kg | Extension - Cohort I Norditropin 0.034 mg/kg | Extension - Cohort I Somapacitan 0.04 mg/kg | Extension - Cohort I Somapacitan 0.08 mg/kg | Extension - Cohort I Somapacitan 0.16 mg/kg | Safety Extension - Cohort I Norditropin 0.034 mg/kg | Safety Extension - Cohort I Somapacitan 0.16 mg/kg | Long Term Safety Extension - Cohort I Norditropin/Somapacitan | Long Term Safety Extension - Cohort I Somapacitan 0.16 mg/kg | Long Term Safety Extension - Cohort II Somapacitan Previously Treated | Long Term Safety Extension - Cohort III Somapacitan Treatment Naive | Long Term Safety Extension - Cohort III Somapacitan Previously Treated | Extension After Week 364 - Cohort I Norditropin/Somapacitan | Extension After Week 364 - Cohort I Somapacitan 0.16 mg/kg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 33
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 16
Not completed — Somapacitan available in their country | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 16

BASELINE CHARACTERISTICS:
Population: Cohort I: full analysis set (FAS) included all randomized participants that received at least one dose of randomized treatment.
  Cohort II and III: All participants enrolled in Cohort II and Cohort III.
Groups:
- Cohort I Norditropin/Somapacitan: Participants received norditropin 0.034 mg/kg subcutaneously daily in main trial period, extension trial period and safety extension trial period. After completing the safety extension trial period (week 156), participants who received norditropin were allocated to open-labelled somapacitan 0.16 mg/kg subcutaneously once weekly for the 104-week safety extension trial period, the 208-week (up till week 364) long-term safety extension period and extension after week 364 period until somapacitan was available for prescription for children with GHD in their country or until August 2024, at the latest.
- Cohort I Somapacitan 0.04 mg/kg: Participants received somapacitan 0.04 mg/kg subcutaneously once-weekly during the 26-week main trial period and the 26-week extension trial period. After completing the main and extension trial periods (week 52), participants received open-labelled somapacitan 0.16 mg/kg/week subcutaneously for the 104-week safety extension trial period, the 208-week (up till week 364) long-term safety extension period and extension after week 364 period until somapacitan was available for prescription for children with GHD in their country or until August 2024, at the latest.
- Cohort I Somapacitan 0.08 mg/kg: Participants received somapacitan 0.08 mg/kg subcutaneously once-weekly during the 26-week main trial period and the 26-week extension trial period. After completing the main and extension trial periods (week 52), participants received open-labelled somapacitan 0.16 mg/kg/week subcutaneously for the 104-week safety extension trial period, the 208-week (up till week 364) long-term safety extension period and extension after week 364 period until somapacitan was available for prescription for children with GHD in their country or until August 2024, at the latest.
- Cohort I Somapacitan 0.16 mg/kg: Participants received somapacitan 0.16 mg/kg subcutaneously once-weekly during the 26-week main trial period and the 26-week extension trial period. After completing the main and extension trial periods (week 52), participants received open-labelled somapacitan 0.16 mg/kg/week subcutaneously for the 104-week safety extension trial period, the 208-week (up till week 364) long-term safety extension period and extension after week 364 period until somapacitan was available for prescription for children with GHD in their country or until August 2024, at the latest.
- Cohort II Somapacitan Previously Treated: Participant who was previously treated with GH prior to enrollment in the trial at week 156, received somapacitan 0.16 mg/kg subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
- Cohort III Somapacitan Treatment Naive: Participants who were naive to treatment with GH prior to enrollment in the trial at week 156, received open-labelled somapacitan 0.16 mg/kg subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
- Cohort III Somapacitan Previously Treated: Participants who were previously treated with GH prior to enrollment in the trial at week 156, received open-labelled somapacitan 0.16 mg/kg subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
- Total: Total of all reporting groups
Arm/Group | Cohort I Norditropin/Somapacitan | Cohort I Somapacitan 0.04 mg/kg | Cohort I Somapacitan 0.08 mg/kg | Cohort I Somapacitan 0.16 mg/kg | Cohort II Somapacitan Previously Treated | Cohort III Somapacitan Treatment Naive | Cohort III Somapacitan Previously Treated | Total
Number analyzed (Participants) | 14 | 16 | 15 | 14 | 1 | 4 | 12 | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.89 (1.98) | 5.61 (1.81) | 5.82 (1.82) | 6.06 (2.32) | 2.5 (0.0) | 12.93 (2.24) | 12.69 (2.02) | 7.25 (3.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 5 | 6 | 0 | 1 | 1 | 25
  Male | 9 | 9 | 10 | 8 | 1 | 3 | 11 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 14 | 15 | 15 | 14 | 1 | 4 | 11 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 8 | 6 | 8 | 1 | 1 | 3 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 7 | 8 | 9 | 6 | 0 | 3 | 9 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity (HV) (cm/Year) During the First 26 Weeks of Treatment, Measured as Standing Height With Stadiometer
Description: Height velocity (HV) was derived from height measurements taken at baseline (week 0) and the week 26 as: HV = (height at 26 weeks visit- height at baseline) / (time from baseline to 26 weeks visit in years).
Time Frame: Baseline (week 0), week 26
Population: FAS was used to analyse this outcome measure. FAS is defined as all randomized participants that received at least one dose of randomized treatment. Here, Overall number of participants analysed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Centimetre per year (Cm/year)
Groups:
- Cohort I - Norditropin 0.034 mg/kg: Participants received norditropin 0.034 mg/kg subcutaneously daily during 26 weeks main trial period.
- Cohort I - Somapacitan 0.04 mg/kg: Participants received somapacitan 0.04 mg/kg subcutaneously once weekly during 26 weeks main trial period.
- Cohort I - Somapacitan 0.08 mg/kg: Participants received somapacitan 0.08 mg/kg subcutaneously once weekly during 26 weeks main trial period.
- Cohort I - Somapcitan 0.16 mg/kg: Participants received somapacitan 0.16 mg/kg subcutaneously once weekly during 26 weeks main trial period.
Arm/Group | Cohort I - Norditropin 0.034 mg/kg | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 14 | 14 | 15 | 14
Centimetre per year (Cm/year) | 11.35 (3.27) | 7.96 (2.04) | 10.92 (1.90) | 12.88 (3.46)
Statistical Analysis 1: Comparison: Cohort I - Norditropin 0.034 mg/kg vs Cohort I - Somapacitan 0.04 mg/kg; The primary analysis tested the estimated treatment difference in HV after 26 weeks of treatment between once-weekly somapacitan 0.04 mg/kg and daily dosing of norditropin 0.034 mg/kg. It was analysed using a mixed model for repeated measurements, with treatment, age group, sex, region and sex by age group interaction as factors and height at baseline as a covariate, all nested within week as a factor; Test type: Other; Estimated Treatment difference = -3.66, 95% CI 2-sided [-5.57 to -1.76]
Statistical Analysis 2: Comparison: Cohort I - Norditropin 0.034 mg/kg vs Cohort I - Somapacitan 0.08 mg/kg; The primary analysis tested the estimated treatment difference in HV after 26 weeks of treatment between once-weekly somapacitan 0.08 mg/kg and daily dosing of norditropin 0.034 mg/kg. It was analysed using a mixed model for repeated measurements, with treatment, age group, sex, region and sex by age group interaction as factors and height at baseline as a covariate, all nested within week as a factor; Test type: Other; Estimated treatment difference = -0.55, 95% CI 2-sided [-2.41 to 1.32]
Statistical Analysis 3: Comparison: Cohort I - Norditropin 0.034 mg/kg vs Cohort I - Somapcitan 0.16 mg/kg; The primary analysis tested the estimated treatment difference in HV after 26 weeks of treatment between once-weekly somapacitan 0.16 mg/kg and daily dosing of norditropin 0.034 mg/kg. It was analysed using a mixed model for repeated measurements, with treatment, age group, sex, region and sex by age group interaction as factors and height at baseline as a covariate, all nested within week as a factor; Test type: Other; Estimated treatment difference = 1.67, 95% CI 2-sided [-0.22 to 3.56]

2. Secondary Outcome: Cohort I: Change in Height Standard Deviation Score (HSDS)
Description: Change in height standard deviation score is presented from baseline (week 0) to end of the main trial period week 26 and end of extension trial period week 52. The formula to calculate HSDS is: HSDS = ((Height / M)**L-1) / (L*S). L: The gender and age-specific power in the Box-Cox transformation, M: The gender and age-specific median, S: The gender and age-specific generalized coefficient of variation. The range for HSDS was -10 to +10. Negative scores indicated a height below the mean height for a child with the same age and gender, whereas positive scores indicated a height above the mean height for a child with the same age and gender.
Time Frame: Baseline (Week 0), week 26, week 52
Population: This outcome measure was assessed only for Cohort 1 and FAS was used to analyse this outcome measure. FAS is defined as all randomised participants that received at least one dose of randomised treatment. Here, Overall number of participants analysed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Cohort I - Norditropin 0.034 mg/kg: Participants received norditropin 0.034 mg/kg subcutaneously daily during 26 weeks main trial period and 26 weeks extension trial period.
- Cohort I - Somapacitan 0.04 mg/kg: Participants received somapacitan 0.04 mg/kg subcutaneously once weekly during 26 weeks main trial period and 26 weeks extension trial period.
- Cohort I - Somapacitan 0.08 mg/kg: Participants received somapacitan 0.08 mg/kg subcutaneously once weekly during 26 weeks main trial period and 26 weeks extension trial period.
- Cohort I - Somapcitan 0.16 mg/kg: Participants received somapacitan 0.16 mg/kg subcutaneously once weekly during 26 weeks main trial period and 26 weeks extension trial period.
Arm/Group | Cohort I - Norditropin 0.034 mg/kg | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 14 | 14 | 15 | 14
Score on scale
  Change at week 26 | 0.66 (0.38) | 0.31 (0.29) | 0.63 (0.29) | 0.89 (0.51)
  Change at week 52 | 0.98 (0.50) | 0.59 (0.46) | 0.95 (0.48) | 1.45 (0.86)

3. Secondary Outcome: Cohort I: Change in Height Velocity Standard Deviation Score (HVSDS)
Description: Change in height velocity standard deviation score is presented from baseline (week 0) to end of main trial period week 26 and end of extension trial period week 52. HVSDS was calculated using the formula: HVSDS = (height velocity - mean)/standard deviation (SD), where height velocity was the height velocity variable measured, mean and SD of height velocity by gender and age for the reference population. The range for HVSDS was -10 to +10. Negative scores indicated a height velocity below the mean height velocity for a child with the same age and gender, whereas positive scores indicated a height velocity above the mean height velocity for a child with the same age and gender.
Time Frame: Baseline (Week 0), week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Cohort I - Norditropin 0.034 mg/kg | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 14 | 14 | 15 | 14
Score on scale
  Change at week 26 | 9.02 (5.03) | 4.93 (3.25) | 7.27 (3.76) | 10.01 (4.67)
  Change at week 52 | 7.41 (4.08) | 4.72 (2.79) | 6.14 (3.36) | 8.60 (3.15)

4. Secondary Outcome: Cohort I: Adverse Events Rate, Including Injection Site Reactions
Description: Adverse events per 100 patient years are presented. AEs with an onset after the first administration of trial product and up until 14 days after last trial drug administration for withdrawn participants, and with an onset after the first administration of trial product and up until visit 32 (week 364) or 14 days after last trial drug administration, which ever comes first, for all other participants, are analysed.
Time Frame: From week 0 Up to week 364
Population: Safety analysis set (SAS) is defined as all randomised participants that received at least one dose of randomised treatment. Data for 3 somapacitan arms (0.04/0.08/0.16 mg/kg) have been pooled from week 156-364, because it was considered appropriate to pool the data from those arms since the size of each individual cohort was small and it would give a more robust measure of long-term safety and tolerability of treatment with somapacitan 0.16 mg/kg/week using this methodology.
Measure: Number; unit: Events per 100 patient years
Groups:
- Cohort I Norditropin 0-156 Week: Participants were randomized to receive norditropin 0.034 mg/kg daily in main trial, extension trial period and open labelled in safety extension trial period.
- Cohort I Norditropin /Somapacitan 0.16 mg/kg Week 156-364: After completing the safety extension trial period (week 156), participants who received norditropin were allocated to open-labelled somapacitan 0.16 mg/kg subcutaneously once weekly for the 208-week (up till week 364) long-term safety extension period.
- Cohort I Somapacitan 0.04 mg/kg Week 0-52: Participants received 0.04 mg/kg subcutaneously once-weekly during the 26 weeks main trial and 26 weeks extension trial period.
- Cohort I Somapacitan 0.08 mg/kg Week 0-52: Participants received 0.08 mg/kg subcutaneously once-weekly during the 26 weeks main trial period and 26 weeks extension trial period.
- Cohort I Somapacitan 0.16 mg/kg Week 0-52: Participants received 0.16 mg/kg subcutaneously once-weekly during the 26 weeks main trial period and 26 weeks extension trial period.
- Cohort I Somapacitan 0.16 mg/kg (Previous Dose 0.04 mg/kg) Week 52-156: Participants initially randomized to double-blinded somapacitan treatment 0.04 mg/kg during main and extension period received open-labelled somapacitan 0.16 mg/kg subcutaneously once-weekly during 104-week safety extension period.
- Cohort I Somapacitan 0.16 mg/kg (Previous Dose 0.08 mg/kg) Week 52-156: Participants initially randomized to double-blinded somapacitan treatment 0.08 mg/kg during main and extension period received open-labelled somapacitan 0.16 mg/kg subcutaneously once-weekly during 104-week safety extension period.
- Cohort I Somapacitan 0.16 mg/kg (Previous Dose 0.16 mg/kg) Week 52-156: Participants initially randomized to double-blinded somapacitan treatment 0.16 mg/kg during main and extension period received open-labelled somapacitan 0.16 mg/kg subcutaneously once-weekly during 104-week safety extension period.
- Cohort I Somapacitan 0.16 mg/kg Week 156 - 364: Participants received somapacitan 0.16 mg/kg subcutaneously once weekly for the 208-week long term safety extension period (up till week 364)
Arm/Group | Cohort I Norditropin 0-156 Week | Cohort I Norditropin /Somapacitan 0.16 mg/kg Week 156-364 | Cohort I Somapacitan 0.04 mg/kg Week 0-52 | Cohort I Somapacitan 0.08 mg/kg Week 0-52 | Cohort I Somapacitan 0.16 mg/kg Week 0-52 | Cohort I Somapacitan 0.16 mg/kg (Previous Dose 0.04 mg/kg) Week 52-156 | Cohort I Somapacitan 0.16 mg/kg (Previous Dose 0.08 mg/kg) Week 52-156 | Cohort I Somapacitan 0.16 mg/kg (Previous Dose 0.16 mg/kg) Week 52-156 | Cohort I Somapacitan 0.16 mg/kg Week 156 - 364
Number analyzed (Participants) | 14 | 11 | 16 | 15 | 14 | 15 | 15 | 14 | 39
Events per 100 patient years | 247.7 | 116.3 | 210.4 | 311.5 | 364.8 | 163.1 | 281.2 | 264.9 | 186.3

5. Secondary Outcome: Cohort I: Occurrence of Anti-NNC0195-0092 and Anti-hGH Antibodies
Description: Participants who developed anti-NNC0195-0092 and anti-hGH antibodies are reported in this outcome measure.
Time Frame: From week 0 Up to week 364
Population: This outcome measure was assessed only for Cohort 1 and SAS was used to analyse this outcome measure. SAS is defined as all randomized participants that received at least one dose of randomized treatment.
  Participants who were randomised to somapacitan 0.04/0.08/0.16 mg/kg/week) received respective doses from week 0 to week 52. From week 52 to week 364, all randomised participants received open labelled somapacitan 0.16 mg/kg/week.
Measure: Number; unit: Participants
Groups:
- Cohort I Norditropin/Somapacitan: Participants received norditropin 0.034 mg/kg subcutaneously daily in main trial period (26 weeks), extension trial period (26 weeks) and 104 week safety extension trial period. In long term safety extension period all participants who received norditropin were allocated to open-labelled somapacitan 0.16 mg/kg subcutaneously once weekly for the 208-week long term safety extension period (up till week 364).
- Cohort I Somapacitan 0.04 mg/kg: Participants received somapacitan 0.04 mg/kg subcutaneously once-weekly during 26 week main trial period and 26 week extension trial period.
- Cohort I Somapacitan 0.08 mg/kg: Participants received somapacitan 0.08 mg/kg subcutaneously once-weekly during 26 week main trial period and 26 week extension trial period.
- Cohort I Somapacitan 0.16 mg/kg: Participants received somapacitan 0.16 mg/kg subcutaneously once-weekly during 26 week main trial period and 26 week extension trial period.
- Cohort I Somapacitan 0.16 mg/kg (Week 52-week 364): After completing the main and extension trial periods (week 52), participants who were initially randomized to double-blinded somapacitan (0.04/0.08/0.16 mg/kg/week) received open-labelled somapacitan 0.16 mg/kg/week subcutaneously during safety extension trial period and 208-week (up till week 364) long-term safety extension period.
Arm/Group | Cohort I Norditropin/Somapacitan | Cohort I Somapacitan 0.04 mg/kg | Cohort I Somapacitan 0.08 mg/kg | Cohort I Somapacitan 0.16 mg/kg | Cohort I Somapacitan 0.16 mg/kg (Week 52-week 364)
Number analyzed (Participants) | 14 | 16 | 15 | 14 | 45
Participants
  Anti-NNC0195-0092 antibody | 0 | 2 | 2 | 2 | 6
  Anti-hGH antibody | 1 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change in Insulin-like Growth Factor I (IGF-I) Standard Deviation Score (SDS)
Description: Change in IGF-I SDS is presented from baseline (week 0) to end of main trial period week 26 and end of extension period week 52. The range for IGF-I SDS was from -10 to +10. Negative scores indicated a IGF-I below the mean IGF-I for a child with the same age and gender, whereas positive scores indicated a IGF-I above the mean IGF-I for a child with the same age and gender.
Time Frame: (Week 0), week 26, week 52
Population: This outcome measure was assessed only for Cohort 1 and FAS was used to analyse this outcome measure. FAS is defined as all randomised participants that received at least one dose of randomised treatment. Here, Overall number of participants analysed = participants with available data for this outcome measure. Number analysed = participants analysed for specific category for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Cohort I - Norditropin 0.034 mg/kg | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 14 | 14 | 14 | 14
Score on scale
  Change at week 26 | 1.86 (0.81) | 0.95 (0.55) | 1.99 (1.02) | 3.00 (1.43)
  Change at week 52: number analyzed (Participants) | 14 | 13 | 14 | 14
  Change at week 52 | 1.67 (1.78) | 0.98 (0.67) | 2.05 (1.00) | 3.29 (1.73)

7. Secondary Outcome: Change in Insulin-like Growth Factor Binding Protein 3 (IGFBP-3) Standard Deviation Score (SDS)
Description: Change in IGFBP-3 SDS is presented from baseline (week 0) to end of main trial period week 26 and end of extension trial period week 52. The range for IGFBP-3 SDS was from -10 to +10. Negative scores indicated a IGFBP-3 below the mean IGFBP-3 for a child with the same age and gender, whereas positive scores indicated a IGFBP-3 above the mean IGFBP-3 for a child with the same age and gender.
Time Frame: Baseline (Week 0), week 26, week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Cohort I - Norditropin 0.034 mg/kg | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 14 | 13 | 14 | 14
Score on scale
  Change at week 26 | 1.58 (0.99) | 0.86 (0.73) | 1.59 (1.04) | 1.45 (1.33)
  Change at week 52 | 0.95 (1.88) | 1.05 (0.87) | 1.54 (1.13) | 1.81 (1.39)

8. Primary Outcome: Cohort II and Cohort III - Adverse Events Rate, Including Injection Site Reactions in Children With GHD.
Description: This primary outcome measure was analysed by cohort using descriptive statistics. Adverse event per 100 patient years are presented in this outcome measure.
Time Frame: From week 156 up to week 364
Population: The outcome measure was assessed only for Cohort II and Cohort III. All participants: all adverse events (AEs) with an onset after the first administration of trial product & up until 14 days after last trial drug administration for withdrawn participants, & with an onset after the first administration of trial product & up until visit 32 (week 208) or 14 days after last trial drug administration, which ever comes first for all participants are included in the analysis.
Measure: Number; unit: Events per 100 patient years
Arm/Group | Cohort II Somapacitan Previously Treated | Cohort III Somapacitan Treatment Naive | Cohort III Somapacitan Previously Treated
Number analyzed (Participants) | 1 | 4 | 12
Events per 100 patient years | 1047 | 115.4 | 196.9

9. Secondary Outcome: Height Velocity (HV) (cm/Year) at Weeks 52 (Derived From Standing Height)
Description: HV was derived from height measurements taken at baseline (week 0) and the week 52 as: HV = (height at 52 weeks visit-height at baseline) / (time from baseline to 52 weeks visit in years)
Time Frame: Baseline (week 0); week 52
Population: This outcome measure was assessed only for Cohort 1 and FAS was used to analyse this outcome measure. FAS is defined as all randomized participants that received at least one dose of randomized treatment. Here, Overall number of participants analysed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Cm/year
Arm/Group | Cohort I - Norditropin 0.034 mg/kg | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 14 | 14 | 15 | 14
Cm/year | 9.8 (2.3) | 7.8 (1.8) | 9.7 (1.8) | 11.5 (2.6)

10. Secondary Outcome: Bone Age Progression vs. Chronological Age Ratio
Description: The bone age vs. chronological age ratio is presented at week 52. X-Ray of left hand and wrist, central assessed according to Greulich & Pyle atlas were taken.
Time Frame: At week 52
Population: This outcome measure was assessed only for Cohort 1 and FAS was used to analyse this outcome measure. FAS is defined as all randomized participants that received at least one dose of randomized treatment. Here, Overall number of participants analysed (N) = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort I - Norditropin 0.034 mg/kg | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 14 | 13 | 15 | 13
Ratio | 0.577 (0.176) | 0.570 (0.147) | 0.651 (0.176) | 0.705 (0.207)

11. Secondary Outcome: Serum Somapacitan Concentrations
Description: Serum somapacitan concentrations are presented at week 52.
Time Frame: At week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Ng/mL
Arm/Group | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 14 | 14 | 14
Ng/mL | 18.381 (20.911) | 44.563 (60.922) | 169.320 (212.233)

12. Secondary Outcome: Changes in Emotional Well-being Score, Physical Health Score, Social Well-being Score and Total Score in TRIM-CGHD-O (Treatment Related Impact Measure - Child Growth Hormone Deficiency- Observer)
Description: Change in Treatment Related Impact Measure from baseline (week 0) to week 26 and week 52 were assessed in children with growth hormone deficiency. This outcome measure was assessed using patient reported outcome (PRO) questionnaires with 3 domains, such as emotional well-being score, physical health score, social wellbeing core and total score. The total score was calculated by taking average of each domain. The scale range for each domain and total score was from 0-100 and a lower score indicates a better health state. TRIMCGHD-O was analysed using descriptive statistics.
Time Frame: Baseline (Week 0), week 26, week 52
Population: This outcome measure was assessed only for Cohort 1 and FAS was used to analyse this outcome measure. FAS is defined as all randomized participants that received at least one dose of randomized treatment. Here, Overall number of participants analysed = participants with available data for this outcome measure. Number analysed = participants analysed for specific category for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Cohort I - Norditropin 0.034 mg/kg | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 14 | 14 | 15 | 14
Score on scale
  Physical health score at week 26: number analyzed (Participants) | 13 | 14 | 15 | 14
  Physical health score at week 26 | 4.3 (18.8) | -4.0 (10.3) | -2.8 (27.0) | -11.6 (16.9)
  Physical health score at week 52: number analyzed (Participants) | 13 | 14 | 15 | 14
  Physical health score at week 52 | -1.9 (13.4) | 0.9 (13.8) | -1.0 (20.9) | -6.7 (16.8)
  Emotional well-being score at week 26: number analyzed (Participants) | 12 | 12 | 13 | 13
  Emotional well-being score at week 26 | -3.3 (19.8) | 1.0 (24.9) | 1.1 (22.0) | 2.4 (28.4)
  Emotional well-being score at week 52: number analyzed (Participants) | 11 | 12 | 13 | 13
  Emotional well-being score at week 52 | -5.7 (13.2) | 1.4 (18.7) | -8.0 (22.7) | -12.2 (27.9)
  Social well-being score at week 26: number analyzed (Participants) | 13 | 13 | 15 | 14
  Social well-being score at week 26 | -9.6 (17.5) | 0.6 (20.3) | -8.6 (17.8) | -11.0 (22.7)
  Social well-being score at week 52: number analyzed (Participants) | 14 | 13 | 14 | 13
  Social well-being score at week 52 | -9.5 (23.9) | 4.5 (20.6) | -20.5 (20.4) | -17.9 (21.2)
  Total score at week 26: number analyzed (Participants) | 13 | 13 | 15 | 14
  Total score at week 26 | -4.6 (10.7) | -0.7 (13.6) | -3.9 (16.4) | -5.9 (12.6)
  Total score at week 52: number analyzed (Participants) | 13 | 13 | 15 | 14
  Total score at week 52 | -6.1 (10.2) | 1.8 (13.5) | -9.4 (17.3) | -12.7 (12.3)

13. Secondary Outcome: Total Score of TB-CGHD-O (The Treatment Burden Measure - Child Growth Hormone Deficiency - Observer)
Description: Total score of Treatment Burden Measure (observer) was assessed at week 26 and at week 52 in children with growth hormone deficiency. This outcome measure was assessed using PRO questionnaires. The scale range for total score was from 0-100 and a lower score indicates a better health state.
Time Frame: At week 26, at week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Cohort I - Norditropin 0.034 mg/kg | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 12 | 14 | 15 | 14
Score on scale
  Total score at week 26: number analyzed (Participants) | 12 | 14 | 14 | 14
  Total score at week 26 | 14.8 (16.2) | 14.0 (11.9) | 10.2 (11.0) | 6.8 (8.9)
  Total score at week 52 | 12.3 (13.9) | 13.7 (13.2) | 11.3 (12.3) | 3.9 (8.1)

14. Secondary Outcome: Total Score of TB-CGHD-P (The Treatment Burden Measure - Child Growth Hormone Deficiency - Parent/Guardian)
Description: Total score of Treatment Burden Measure (parent/guardian) is reported at week 26 and at week 52 in children with growth hormone deficiency. This outcome measure was assessed using PRO questionnaires. The scale range for total score was from 0-100 and a lower score indicates a better health state.
Time Frame: At week 26, at week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Cohort I - Norditropin 0.034 mg/kg | Cohort I - Somapacitan 0.04 mg/kg | Cohort I - Somapacitan 0.08 mg/kg | Cohort I - Somapcitan 0.16 mg/kg
Number analyzed (Participants) | 13 | 14 | 15 | 14
Score on scale
  Total score at week 26 | 26.9 (24.7) | 24.6 (16.7) | 17.5 (20.5) | 18.8 (22.2)
  Total score at week 52 | 23.6 (27.3) | 19.6 (19.0) | 13.8 (12.5) | 15.6 (16.6)

ADVERSE EVENTS:
Time Frame: Week 0 to week 442
Description: Cohort I: SAS is defined as all randomised participants that received at least one dose of randomised treatment.
  Cohort II and III: All participants enrolled in Cohort II and Cohort III.
  All presented AEs are TEAEs (treatment emergent adverse events). Adverse events will be defined as "treatment-emergent", if the onset of the event occurs in the on-treatment period.
Groups:
- Cohort I - Norditropin (Week 0-156): Participants were randomized to receive norditropin 0.034 mg/kg daily in main trial, extension trial period and open labelled in safety extension trial period.
- Cohort I - Norditropin/Somapacitan 0.16 mg/kg (Week 156-364): After completing the safety extension trial period (week 156), participants who received norditropin were allocated to open-labelled somapacitan 0.16 mg/kg subcutaneously once weekly for the 208-week (up till week 364) long-term safety extension period.
- Cohort I - Norditropin/Somapacitan 0.16 mg/kg (Week >364): Participants received somapacitan 0.16 mg/kg subcutaneously once weekly from week 364 until somapacitan was available for prescription for children with GHD in their country or until August 2024, at the latest.
- Cohort I - Somapacitan 0.04 mg/kg (Week 0-52): Participants received somapacitan 0.04 mg/kg subcutaneously once weekly during 26 weeks main trial period and 26 weeks extension trial period.
- Cohort I - Somapacitan 0.08 mg/kg (Week 0-52): Participants received somapacitan 0.08 mg/kg subcutaneously once weekly during 26 weeks main trial period and 26 weeks extension trial period.
- Cohort I - Somapacitan 0.16 mg/kg (Week 0-52): Participants received somapacitan 0.16 mg/kg subcutaneously once weekly during 26 weeks main trial period and 26 weeks extension trial period.
- Cohort I - Somapacitan 0.16 mg/kg (Week 52-442): After completing the main and extension trial periods (week 52), participants who were initially randomized to double-blinded somapacitan (0.04/0.08/0.16 mg/kg/week) received open-labelled somapacitan 0.16 mg/kg/week subcutaneously during safety extension trial period, 208-week (up till week 364) long-term safety extension period and until somapacitan was available for prescription for children with GHD in their country or until August 2024, at the latest.
- Cohort II - Somapacitan (0.16 mg/kg) Previously Treated: Participant who was previously treated with GH prior to enrollment in the trial at week 156, received somapacitan 0.16 mg/kg subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
- Cohort III - Somapacitan (0.16 mg/kg) Treatment Naive: Participants who were naive to treatment with GH prior to enrollment in the trial at week 156, received open-labelled somapacitan 0.16 mg/kg subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
- Cohort III - Somapacitan (0.16 mg/kg) Previously Treated: Participants who were previously treated with GH prior to enrollment in the trial at week 156, received open-labelled somapacitan 0.16 mg/kg subcutaneously once weekly until it was available for prescription in participants' respective countries or until August 2024, at the latest.
Arm/Group | Cohort I - Norditropin (Week 0-156) | Cohort I - Norditropin/Somapacitan 0.16 mg/kg (Week 156-364) | Cohort I - Norditropin/Somapacitan 0.16 mg/kg (Week >364) | Cohort I - Somapacitan 0.04 mg/kg (Week 0-52) | Cohort I - Somapacitan 0.08 mg/kg (Week 0-52) | Cohort I - Somapacitan 0.16 mg/kg (Week 0-52) | Cohort I - Somapacitan 0.16 mg/kg (Week 52-442) | Cohort II - Somapacitan (0.16 mg/kg) Previously Treated | Cohort III - Somapacitan (0.16 mg/kg) Treatment Naive | Cohort III - Somapacitan (0.16 mg/kg) Previously Treated
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11 | 0/5 | 0/16 | 0/15 | 0/14 | 0/44 | 0/1 | 0/4 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/11 | 0/5 | 0/16 | 1/15 | 1/14 | 6/44 | 1/1 | 0/4 | 0/12
Other Adverse Events (participants affected / at risk) | 14/14 | 10/11 | 2/5 | 11/16 | 11/15 | 13/14 | 35/44 | 1/1 | 2/4 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I - Norditropin (Week 0-156) (N=14) | Cohort I - Norditropin/Somapacitan 0.16 mg/kg (Week 156-364) (N=11) | Cohort I - Norditropin/Somapacitan 0.16 mg/kg (Week >364) (N=5) | Cohort I - Somapacitan 0.04 mg/kg (Week 0-52) (N=16) | Cohort I - Somapacitan 0.08 mg/kg (Week 0-52) (N=15) | Cohort I - Somapacitan 0.16 mg/kg (Week 0-52) (N=14) | Cohort I - Somapacitan 0.16 mg/kg (Week 52-442) (N=44) | Cohort II - Somapacitan (0.16 mg/kg) Previously Treated (N=1) | Cohort III - Somapacitan (0.16 mg/kg) Treatment Naive (N=4) | Cohort III - Somapacitan (0.16 mg/kg) Previously Treated (N=12)
Adenoidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I - Norditropin (Week 0-156) (N=14) | Cohort I - Norditropin/Somapacitan 0.16 mg/kg (Week 156-364) (N=11) | Cohort I - Norditropin/Somapacitan 0.16 mg/kg (Week >364) (N=5) | Cohort I - Somapacitan 0.04 mg/kg (Week 0-52) (N=16) | Cohort I - Somapacitan 0.08 mg/kg (Week 0-52) (N=15) | Cohort I - Somapacitan 0.16 mg/kg (Week 0-52) (N=14) | Cohort I - Somapacitan 0.16 mg/kg (Week 52-442) (N=44) | Cohort II - Somapacitan (0.16 mg/kg) Previously Treated (N=1) | Cohort III - Somapacitan (0.16 mg/kg) Treatment Naive (N=4) | Cohort III - Somapacitan (0.16 mg/kg) Previously Treated (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anisometropia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Autism spectrum disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (17) | 1 (1) | 1 (1) | 3 (4)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Cranial operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 2 (5) | 1 (2) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Educational problem (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (9) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 1 (1) | 2 (3)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 9 (14) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Microcytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mumps (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (12) | 2 (4) | 0 (0) | 0 (0) | 1 (7) | 3 (8) | 8 (52) | 1 (12) | 1 (1) | 3 (8)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic nerve cupping (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 6 (8) | 1 (7) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 1 (4)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (5) | 1 (6) | 0 (0) | 6 (8) | 1 (1) | 1 (1) | 12 (20) | 1 (5) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (11) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensory processing disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Social problem (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Speech disorder developmental (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (22) | 0 (0) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (6) | 1 (4) | 0 (0) | 3 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3)
Varicella (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 0 (0) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dientamoeba infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematology test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property"

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT02616562/Prot_SAP_000.pdf